CLINICAL TRIAL: NCT02817698
Title: Imaging the Neurochemistry of Drug Addiction With PET
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kelly Cosgrove, Associate Professor, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1604017594; 1R01DA038709-01A1 (NIH); 1R01DA038832-01A1 (NIH); 1R03DA047588-01 (NIH)
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Smoking; Cannabis
Keywords: smoking; cannabis; cocaine
MeSH Terms: conditions — Smoking; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug of dependence (Experimental): There is only one arm to the study. All subjects will receive their drug of dependence in this study. Nicotine dependent subjects will receive tobacco cigarettes, cannabis dependent subjects will receive cannabis cigarettes, and cocaine dependent subjects will receive IV cocaine.
  Interventions: Drug: cannabis

INTERVENTIONS:
Drug: cannabis — All cannabis dependent subjects will use cannabis cigarettes to induce elevated dopamine and beta endorphin levels in the brain.
  Other Names: marijuana

SUMMARY:
The investigators' project has two overarching goals. 1) The investigators will use newly developed positron emission tomography (PET) technology to investigate the dopaminergic neurochemistry of drugs of abuse including marijuana, traditional cigarettes, and cocaine, and 2) The investigators will extend PET technology to an additional neurotransmitter system - namely, the opioid-ergic system, using the same drugs of abuse.

DETAILED DESCRIPTION:
Aim 1. To examine the magnitude, location and timing of drug-induced dopamine release.

1. Tobacco smokers (n=20) will be imaged with [11C]raclopride PET, after overnight abstinence from tobacco. Subjects will smoke their preferred brand of cigarette during the PET scan.
2. Marijuana smokers (n=20) will be imaged with [11C]raclopride PET, after overnight abstinence from marijuana. Subjects will smoke a marijuana cigarette during the PET scan.
3. Cocaine users (n=20) will be imaged with [11C]raclopride PET, after overnight abstinence from cocaine. Subjects will be administered cocaine during the PET scan.

Aim 2. To examine the magnitude, location and timing of drug-induced beta-endorphin release. *The Investigators will attempt to use the same subjects from Aim 1 for Aim 2.

1. Tobacco smokers (n=20) will be imaged with [11C]carfentanil PET, after overnight abstinence from tobacco. Subjects will smoke their preferred brand of cigarette during the PET scan.
2. Marijuana smokers (n=20) will be imaged with [11C]carfentanil PET, after overnight abstinence from marijuana. Subjects will smoke a marijuana cigarette during the PET scan.
3. Cocaine users (n=20) will be imaged with [11C]carfentanil PET, after overnight abstinence from cocaine. Subjects will be administered cocaine during the PET scan.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria:

  1. Men and women, aged 18-55 years
  2. Able to read and write English and give voluntary written informed consent
  3. Not treatment seeking or using treatment medications

Tobacco Smokers

1. Have a Fagerström Test for Nicotine Dependence (FTND) rating of at least 3.
2. Have been using at least 7 cigarettes per day for at least 1 year
3. Carbon monoxide levels > 10 ppm during intake evaluation
4. Urine cotinine levels of > 150 ng/mL during intake evaluation
5. Are not current users of marijuana or other illicit drugs

Marijuana Smokers

1. Meet DSM-V criteria for cannabis use disorder based on the structured clinical interview diagnostic (SCID) or regular cannabis use of >5 times/week
2. Test positive for THC
3. Have been smoking cannabis on a regular basis for > 1 year

Cocaine Users

1. DSM-V criteria for Cocaine Abuse or Dependence
2. Recent street cocaine use in excess of amounts to be administered in the current study
3. Intravenous and/or smoked (crack/ freebase) use
4. Positive urine toxicology screen for cocaine

Exclusion Criteria:

* 1. Current significant medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology.

  2. History of or current neurological or significant psychiatric disorder such as schizophrenia or bipolar disorder (DSM-IV Axis 1).

  3. History of significant head trauma. 4. Women who are pregnant or nursing, or fail to use one of the following methods of birth control unless she or partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or IUD).

  5. Regular or current significant use of any prescription, herbal or illegal psychotropic medications (e.g., antidepressants, antipsychotics, anxiolytics, ecstasy) in the past 6 mo, with no current illegal drug use confirmed by urine toxicology (except for cocaine and marijuana when relevant).

  6. Significant substance misuse (including alcohol, and excluding cannabis and marijuana when relevant) that in the PI's determination interferes with the study results or safety of the subject.

  7. Have MRI-incompatible implants and other contraindications for MRI, such as a pacemaker, artificial joints, non-removable body piercings, claustrophobia, etc.

  8. Subjects with history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over FDA limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year.

  9. Subjects with current, past or anticipated exposure to radiation in the work place within one year of proposed research PET scans.

  10. Subjects with history of IV drug use which would prevent venous access for PET tracer injection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2024-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Cosgrove, PhD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Connecticut Mental Health Center, New Haven, Connecticut
  - Yale Magnetic Resonance Research Center, New Haven, Connecticut
  - Yale PET Center, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Calakos KC, Liu H, Lu Y, Anderson JM, Matuskey D, Nabulsi N, Ye Y, Skosnik PD, D'Souza DC, Morris ED, Cosgrove KP, Hillmer AT. Assessment of transient dopamine responses to smoked cannabis. Drug Alcohol Depend. 2021 Oct 1;227:108920. doi: 10.1016/j.drugalcdep.2021.108920. Epub 2021 Jul 29. PMID 34399137

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug of Dependence
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Drug of Dependence
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 29.52 [19 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Dopamine Levels at Baseline and After Drug of Dependence Administration as Confirmed by PET Images.
Description: PET images will be obtained in dependent subjects at baseline and after drug of dependence administration. Change in DA levels will be determined by change in binding potential of raclopride. Baseline levels will be assessed during the first scan in the morning after overnight abstinence from their drug of dependence using a 90-minute PET acquisition. Then, drug of dependence will be administered 35 minutes before a second 90-minute PET acquisition. The beginning of the second PET scan will be approximately 5 hours after the beginning of the first PET scan, however in some cases this may be longer, or the scans may take place on separate days due to scheduling constraints or scan cancellations.
Time Frame: 90 minute PET scan acquisition. Drug of dependence will be given at -35 mins
Population: Subjects were analyzed based on cluster size with a threshold of 16 voxels.
Measure: Mean (Full Range); unit: mm^3
Arm/Group | Drug of Dependence
Number analyzed (Participants) | 12
mm^3
  R VS: number analyzed (Participants) | 10
  R VS | 0.0388 [0.022 to 0.058]
  R Putamen: number analyzed (Participants) | 4
  R Putamen | 0.033 [0.028 to 0.038]
  R Caudate: number analyzed (Participants) | 2
  R Caudate | 0.0285 [0.027 to 0.03]
  L VS: number analyzed (Participants) | 5
  L VS | 0.0368 [0.025 to 0.052]
  L Caudate: number analyzed (Participants) | 2
  L Caudate | 0.038 [0.035 to 0.041]
  R VS/Caudate: number analyzed (Participants) | 1
  R VS/Caudate | 0.035 [0.035 to 0.035]
  L Putamen: number analyzed (Participants) | 2
  L Putamen | 0.037 [0.022 to 0.052]

2. Primary Outcome: Change in Beta Endorphin Levels at Baseline and After Drug of Dependence Administration as Confirmed by PET Images.
Description: PET images will be obtained in dependent subjects at baseline and after drug of dependence administration. Change in beta endorphin levels will be determined by change in binding potential of carfentanil. Baseline levels will be assessed during the first scan in the morning after 12 hour abstinence from their drug of dependence using a 90-minute PET acquisition. Then, drug of dependence will be administered 35 minutes before a second 90-minute PET acquisition. The beginning of the second PET scan will be approximately 5 hours after the beginning of the first PET scan, however in some cases this may be longer, or the scans may take place on separate days due to scheduling constraints or scan cancellations.
Time Frame: 120 minute PET scan acquisition. Drug of dependence will be given at -35 mins
Measure: Mean (Full Range); unit: mm^3
Arm/Group | Drug of Dependence
Number analyzed (Participants) | 8
mm^3
  Front | -0.0068 [-0.0501 to 0.0237]
  Amygdala | 0.0190 [-0.2803 to 0.3490]
  Thalamus | 0.0146 [-0.0355 to 0.0748]
  Caudate | 0.0082 [-0.1278 to 0.1310]
  Putamen | 0.0100 [-0.0342 to 0.0865]
  Cingulum | 0.0233 [-0.0687 to 0.0909]
  Insula | 0.0153 [-0.0432 to 0.0910]

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Drug of Dependence
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 1/25
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug of Dependence (N=25)
Anxiety/Tachycardia (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT02817698/Prot_SAP_000.pdf